CLINICAL TRIAL: NCT00373958
Title: A Phase 3, Randomized, Active-Controlled, Double-blind Trial Evaluating the Safety, Tolerability and Immunologic Noninferiority of a 13-valent Pneumococcal Conjugate Vaccine Compared to a 7-valent Pneumococcal Conjugate Vaccine in Healthy Infants Given With Routine Pediatric Vaccinations in the United States
Brief Title: Study Comparing 13-valent Pneumococcal Conjugate Vaccine With 7-valent Pneumococcal Conjugate Vaccine
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Pfizer (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: 6096A1-004
Record Dates: First submitted 2006-09-07; First posted 2006-09-08 (Estimated); Results first posted 2013-02-21 (Estimated); Last update posted 2013-02-21 (Estimated); Status verified 2013-01

CONDITIONS: Vaccines, Pneumococcal

ARMS (2):
- 13vPnC vaccine (Experimental)
  Interventions: Biological: 13 valent pneumococcal conjugate vaccine
- 7vPnC vaccine (Active Comparator)
  Interventions: Biological: 7vPnc pneumococcal conjugate vaccine

INTERVENTIONS:
Biological: 13 valent pneumococcal conjugate vaccine — 1 single 0.5 mL dose together with a concomitant dose of Pediarix and ActHIB at the 2-, 4-, and 6-month visits and ProQuad, PedvaxHIB, and VAQTA at the 12-15 month visit.
  Arms: 13vPnC vaccine
Biological: 7vPnc pneumococcal conjugate vaccine — 1 single 0.5 mL dose together with a concomitant dose of Pediarix and ActHIB at the 2-, 4-, and 6-month visits and ProQuad, PedvaxHIB, and VAQTA at the 12-15 month visit.
  Arms: 7vPnC vaccine

SUMMARY:
The purpose of this study is to evaluate the safety, tolerability, and immunogenicity of the 13-valent pneumococcal vaccine (13vPnC) compare to the 7-valent pneumococcal vaccine (7vPnC) and to compare the immune response to concomitant vaccines administered with 13vPnC and 7vPnC.

ELIGIBILITY:
Inclusion Criteria:

* Healthy 2-month-old infants.
* Available for the entire study period.

Exclusion criteria:

* Previous vaccination with any vaccine before the start of the study.
* Known contraindication to vaccination.

Ages: 42 Days to 98 Days | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 666 (Actual)
Dates: Start 2006-09; Primary Completion 2008-06 (Actual); Study Completion 2008-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Medical Monitor, Study Director — Wyeth is now a wholly owned subsidiary of Pfizer
Locations (34):
- United States (34):
  - Fayetteville, Arkansas
  - Jonesboro, Arkansas
  - Little Rock, Arkansas
  - Downey, California
  - Fontana, California
  - Loma Linda, California
  - Paramount, California
  - Riverside, California
  - Centennial, Colorado
  - Norwich, Connecticut
  - Tampa, Florida
  - Marietta, Georgia
  - Woodstock, Georgia
  - Chicago, Illinois
  - Park Ridge, Illinois
  - Overland Park, Kansas
  - Bardstown, Kentucky
  - Louisville, Kentucky
  - Rochester, New York
  - The Bronx, New York
  - Cincinnati, Ohio
  - Cleveland, Ohio
  - Mason, Ohio
  - Latrobe, Pennsylvania
  - Pittsburgh, Pennsylvania
  - Sellersville, Pennsylvania
  - Wexford, Pennsylvania
  - Charleston, South Carolina
  - Jackson, Tennessee
  - The Woodlands, Texas
  - Murray, Utah
  - Provo, Utah
  - Richmond, Virginia
  - Vienna, Virginia

REFERENCES:
- [Derived] Bryant KA, Gurtman A, Girgenti D, Reisinger K, Johnson A, Pride MW, Patterson S, Devlin C, Gruber WC, Emini EA, Scott DA. Antibody responses to routine pediatric vaccines administered with 13-valent pneumococcal conjugate vaccine. Pediatr Infect Dis J. 2013 Apr;32(4):383-8. doi: 10.1097/INF.0b013e318279e9a9. PMID 23104129
- [Derived] Yeh SH, Gurtman A, Hurley DC, Block SL, Schwartz RH, Patterson S, Jansen KU, Love J, Gruber WC, Emini EA, Scott DA; 004 Study Group. Immunogenicity and safety of 13-valent pneumococcal conjugate vaccine in infants and toddlers. Pediatrics. 2010 Sep;126(3):e493-505. doi: 10.1542/peds.2009-3027. Epub 2010 Aug 23. PMID 20732948

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants were recruited in the United States from September 2006 to January 2008.
Pre-assignment Details: Participants were enrolled into the study according to inclusion/exclusion criteria without a screening period.
Groups:
- 13vPnC: Participants received one single 0.5 mL dose of 13-valent pneumococcal conjugate vaccine (13vPnC) coadministered with Haemophilus b Conjugate Vaccine (ActHIB) and Diphtheria and Tetanus Toxoids and Acellular Pertussis Adsorbed, Hepatitis B (Recombinant) and Inactivated Poliovirus Vaccine Combined (Pediarix) at 2, 4, 6 months (infant series). Participants received one single 0.5 mL dose of 13vPnC coadministered with measles, mumps, rubella varicella vaccine live (ProQuad), Haemophilus b Conjugate Vaccine (Meningococcal Protein Conjugate) (PedvaxHIB), and Hepatitis A Vaccine, Inactivated (VAQTA) at 12-15 months of age (toddler dose).
- 7vPnC: Participants received one single 0.5 mL dose of 7-valent pneumococcal conjugate vaccine (7vPnC) coadministered with Haemophilus b Conjugate Vaccine (ActHIB) and Diphtheria and Tetanus Toxoids and Acellular Pertussis Adsorbed, Hepatitis B (Recombinant) and Inactivated Poliovirus Vaccine Combined (Pediarix) at 2, 4, 6 months (infant series). Participants received one single 0.5 mL dose of 7vPnC coadministered with measles, mumps, rubella varicella vaccine live (ProQuad), Haemophilus b Conjugate Vaccine (Meningococcal Protein Conjugate) (PedvaxHIB), and Hepatitis A Vaccine, Inactivated (VAQTA) at 12-15 months of age (toddler dose).
Period: Infant Series
Arm/Group | 13vPnC | 7vPnC
Started | 334 (One participant was prerandomized but not consented.) | 332
Vaccinated Dose 1 | 332 | 331
Vaccinated Dose 2 | 309 | 305
Vaccinated Dose 3 | 298 | 300
Completed | 294 | 290
Not Completed | 40 | 42
Not completed — Withdrawal by Subject | 13 | 15
Not completed — Failed to return | 8 | 13
Not completed — Lost to Follow-up | 6 | 5
Not completed — Protocol Violation | 3 | 7
Not completed — Lost Kaiser coverage | 4 | 0
Not completed — Child relocated | 1 | 0
Not completed — Consent was not received | 1 | 0
Not completed — Adverse Event | 3 | 1
Not completed — Physician Decision | 1 | 1
Period: Toddler Dose
Arm/Group | 13vPnC | 7vPnC
Started | 294 | 290
Withdrawn After Infant Series | 22 | 25
Vaccinated Toddler Dose | 272 | 265
Completed | 264 | 252
Not Completed | 30 | 38
Not completed — Lost to Follow-up | 5 | 8
Not completed — Withdrawal by Subject | 2 | 2
Not completed — Failed to return | 1 | 2
Not completed — Protocol Violation | 0 | 1
Not completed — Withdrawn after infant series | 22 | 25

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | 13vPnC | 7vPnC | Total
Number analyzed (Participants) | 334 | 332 | 666
Age Continuous [Mean (Standard Deviation); unit: months] | 2.1 (0.3) | 2.1 (0.3) | 2.1 (0.3)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 165 | 139 | 304
  Male | 169 | 193 | 362

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Participants Achieving Antibody Level ≥0.35 μg/mL in 13vPnC Group Relative to 7vPnC Group After the 3-Dose Infant Series
Description: Percentages of Participants achieving World Health Organization (WHO) predefined antibody threshold ≥0.35 μg/mL along with the corresponding 95% CI for the 7 common pneumococcal serotypes (serotypes 4, 6B, 9V, 14, 18C, 19F, and 23F) and 6 additional pneumococcal serotypes specific to 13vPnC (serotypes 1, 3, 5, 6A, 7F, and 19A) are presented.
Time Frame: One month after the 3-dose infant series (7 months of age)
Population: Evaluable immunogenicity (per protocol) population consisting of participants who adhered to the protocol requirements, had valid and determinate assay results, and had no other major protocol violations; (n) = number of participants with a determinate IgG antibody concentration to the given serotype.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | 13vPnC | 7vPnC
Number analyzed (Participants) | 252 | 252
percentage of participants
  Common Serotypes - Serotype 4 (n=252,251) | 94.4 [90.9 to 96.9] | 98.0 [95.4 to 99.4]
  Common Serotypes - Serotype 6B (n=252,250) | 87.3 [82.5 to 91.1] | 92.8 [88.9 to 95.7]
  Common Serotypes - Serotype 9V (n=252,252) | 90.5 [86.2 to 93.8] | 98.4 [96.0 to 99.6]
  Common Serotypes - Serotype 14 (n=251,252) | 97.6 [94.9 to 99.1] | 97.2 [94.4 to 98.9]
  Common Serotypes - Serotype 18C (n=252,252) | 96.8 [93.8 to 98.6] | 98.4 [96.0 to 99.6]
  Common Serotypes - Serotype 19F (n=252,251) | 98.0 [95.4 to 99.4] | 97.6 [94.9 to 99.1]
  Common Serotypes - Serotype 23F (n=252,252) | 90.5 [86.2 to 93.8] | 94.0 [90.4 to 96.6]
  Additional Serotypes - Serotype 1 (n=252,248) | 95.6 [92.3 to 97.8] | 1.6 [0.4 to 4.1]
  Additional Serotypes - Serotype 3 (n=249,241) | 63.5 [57.1 to 69.4] | 4.6 [2.3 to 8.0]
  Additional Serotypes - Serotype 5 (n=252,197) | 89.7 [85.2 to 93.1] | 31.0 [24.6 to 37.9]
  Additional Serotypes - Serotype 6A (n=252,240) | 96.0 [92.8 to 98.1] | 42.5 [36.2 to 49.0]
  Additional Serotypes - Serotype 7F (n=252,248) | 98.4 [96.0 to 99.6] | 2.8 [1.1 to 5.7]
  Additional Serotypes - Serotype 19A (n=251,238) | 98.4 [96.0 to 99.6] | 86.6 [81.6 to 90.6]
Statistical Analysis 1: Comparison: 13vPnC vs 7vPnC; For serotype 4 the difference in percentages between the two groups (13vPnC - 7vPnC) was calculated; Test type: Non-Inferiority or Equivalence — Non-inferiority for each common serotype was declared if the lower limit of the 2-sided 95% CI for the difference between the 2 groups > -10%; Difference = -3.6, 95% CI [-7.3 to -0.1]
Statistical Analysis 2: Comparison: 13vPnC vs 7vPnC; For serotype 6B the difference in percentages between the two groups (13vPnC - 7vPnC) was calculated; Test type: Non-Inferiority or Equivalence — [test comment as in outcome 1, analysis 1]; Difference = -5.5, 95% CI [-10.9 to -0.1]
Statistical Analysis 3: Comparison: 13vPnC vs 7vPnC; For serotype 9V the difference in percentages between the two groups (13vPnC - 7vPnC) was calculated; Test type: Non-Inferiority or Equivalence — [test comment as in outcome 1, analysis 1]; Difference = -7.9, 95% CI [-12.4 to -4.0]
Statistical Analysis 4: Comparison: 13vPnC vs 7vPnC; For serotype 14 the difference in percentages between the two groups (13vPnC - 7vPnC) was calculated; Test type: Non-Inferiority or Equivalence — [test comment as in outcome 1, analysis 1]; Difference = 0.4, 95% CI [-2.7 to 3.5]
Statistical Analysis 5: Comparison: 13vPnC vs 7vPnC; For serotype 18C the difference in percentages between the two groups (13vPnC - 7vPnC) was calculated; Test type: Non-Inferiority or Equivalence — [test comment as in outcome 1, analysis 1]; Difference = -1.6, 95% CI [-4.7 to 1.2]
Statistical Analysis 6: Comparison: 13vPnC vs 7vPnC; For serotype 19F the difference in percentages between the two groups (13vPnC - 7vPnC) was calculated; Test type: Non-Inferiority or Equivalence — [test comment as in outcome 1, analysis 1]; Difference = 0.4, 95% CI [-2.4 to 3.4]
Statistical Analysis 7: Comparison: 13vPnC vs 7vPnC; For serotype 23F the difference in percentages between the two groups (13vPnC - 7vPnC) was calculated; Test type: Non-Inferiority or Equivalence — [test comment as in outcome 1, analysis 1]; Difference = -3.6, 95% CI [-8.5 to 1.2]

2. Primary Outcome: Geometric Mean Antibody Concentration in 13vPnC Group Relative to 7vPnC Group 1 Month After the Toddler Dose
Description: Antibody concentration/geometric mean concentration as measured by enzyme-linked immunosorbent assay (ELISA) for 7 common pneumococcal serotypes (serotypes 4, 6B, 9V, 14, 18C, 19F, and 23F) and 6 additional pneumococcal serotypes specific to 13vPnC (Serotypes 1, 3, 5, 6A, 7F, and 19A) are presented.
Time Frame: 1 Month After the Toddler Dose
Population: Evaluable immunogenicity (per protocol) population of eligible participants, had valid and determinate assay results, and had no other major protocol violations; (n) = number of participants with a determinate antibody concentration for the specified serotype.
Measure: Geometric Mean (95% Confidence Interval); unit: μg/mL
Arm/Group | 13vPnC | 7vPnC
Number analyzed (Participants) | 239 | 223
μg/mL
  Common Serotypes - Serotype 4 (n=235,223) | 3.73 [3.28 to 4.24] | 5.49 [4.91 to 6.13]
  Common Serotypes - Serotype 6B (n=234,223) | 11.53 [9.99 to 13.30] | 15.63 [13.80 to 17.69]
  Common Serotypes - Serotype 9V (n=234,223) | 2.62 [2.32 to 2.94] | 3.63 [3.25 to 4.05]
  Common Serotypes - Serotype 14 (n=235,223) | 9.11 [7.95 to 10.45] | 12.72 [11.22 to 14.41]
  Common Serotypes - Serotype 18C (n=236,223) | 3.20 [2.82 to 3.64] | 4.70 [4.18 to 5.28]
  Common Serotypes - Serotype 19F (n=235,223) | 6.60 [5.85 to 7.44] | 5.60 [4.87 to 6.43]
  Common Serotypes - Serotype 23F (n=234,222) | 5.07 [4.41 to 5.83] | 7.84 [6.91 to 8.90]
  Additional Serotypes - Serotype 1 (n=235,223) | 5.06 [4.43 to 5.80] | 0.03 [0.03 to 0.03]
  Additional Serotypes - Serotype 3 (n=232,223) | 0.94 [0.83 to 1.05] | 0.07 [0.05 to 0.08]
  Additional Serotypes - Serotype 5 (n=235,223) | 3.72 [3.31 to 4.18] | 0.55 [0.47 to 0.64]
  Additional Serotypes - Serotype 6A (n=235,223) | 8.20 [7.30 to 9.20] | 1.87 [1.60 to 2.19]
  Additional Serotypes - Serotype 7F (n=235,223) | 5.67 [5.01 to 6.42] | 0.05 [0.04 to 0.05]
  Additional Serotypes - Serotype 19A (n=236,223) | 8.55 [7.64 to 9.56] | 3.54 [3.15 to 3.98]
Statistical Analysis 1: Comparison: 13vPnC vs 7vPnC; For serotype 4 the GMC ratio (13vPnC/7vPnC) was calculated; Test type: Non-Inferiority or Equivalence — Non-inferiority for each common serotype was declared if the lower limit of the 2-sided 95% CI for the GMC ratio (13vPnC/7vPnC) > 0.5 (2-fold criterion); Ratio = 0.68, 95% CI [0.57 to 0.80]
Statistical Analysis 2: Comparison: 13vPnC vs 7vPnC; For serotype 6B the GMC ratio (13vPnC/7vPnC) was calculated; Test type: Non-Inferiority or Equivalence — [test comment as in outcome 2, analysis 1]; Ratio = 0.74, 95% CI [0.61 to 0.89]
Statistical Analysis 3: Comparison: 13vPnC vs 7vPnC; For serotype 9V the GMC ratio (13vPnC/7vPnC) was calculated; Test type: Non-Inferiority or Equivalence — [test comment as in outcome 2, analysis 1]; Ratio = 0.72, 95% CI [0.62 to 0.85]
Statistical Analysis 4: Comparison: 13vPnC vs 7vPnC; For serotype 14 the GMC ratio (13vPnC/7vPnC) was calculated; Test type: Non-Inferiority or Equivalence — [test comment as in outcome 2, analysis 1]; Ratio = 0.72, 95% CI [0.60 to 0.86]
Statistical Analysis 5: Comparison: 13vPnC vs 7vPnC; For serotype 18C the GMC ratio (13vPnC/7vPnC) was calculated; Test type: Non-Inferiority or Equivalence — [test comment as in outcome 2, analysis 1]; Ratio = 0.68, 95% CI [0.57 to 0.81]
Statistical Analysis 6: Comparison: 13vPnC vs 7vPnC; For serotype 19F the GMC ratio (13vPnC/7vPnC) was calculated; Test type: Non-Inferiority or Equivalence — [test comment as in outcome 2, analysis 1]; Ratio = 1.18, 95% CI [0.98 to 1.41]
Statistical Analysis 7: Comparison: 13vPnC vs 7vPnC; For serotype 23F the GMC ratio (13vPnC/7vPnC) was calculated; Test type: Non-Inferiority or Equivalence — [test comment as in outcome 2, analysis 1]; Ratio = 0.65, 95% CI [0.54 to 0.78]

3. Primary Outcome: Percentage of Participants Achieving Predefined Antibody Levels for Haemophilus Influenzae Type b, Diphtheria Toxoid, and Pertussis Antigens in 13vPnC Group Relative to 7vPnC Group After the Infant Series
Description: Predefined Antibody Levels for Haemophilus Influenzae Type b ([Hib] 0.15 µg/mL or 1.0 µg/mL), Diphtheria Toxoid (0.1 International Units [IU]/mL), and Pertussis antigens (Pertussis filamentous hemagglutinin [FHA] 40.5 Elisa Units [EU]/mL, Pertussis toxoid [PT] 16.5 EU/mL, Pertussis pertactin [PRN] 26 EU/mL).
Time Frame: One Month After the Infant Series (7 months of age)
Population: Evaluable immunogenicity (per protocol) population who adhered to the protocol requirements, had valid and determinate assay results, and had no other major protocol violations. (n) = number of participants with a determinate postinfant series antibody concentration to the given concomitant antigen.
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | 13vPnC | 7vPnC
Number analyzed (Participants) | 252 | 252
Percentage of participants
  Hib 0.15 µg/mL (n=237,230) | 97.9 [95.1 to 99.3] | 97.8 [95.0 to 99.3]
  Hib 1.0 µg/mL (n=237,230) | 77.6 [71.8 to 82.8] | 78.3 [72.4 to 83.4]
  Diphtheria [IU]/mL (n=233,230) | 95.7 [92.2 to 97.9] | 96.1 [92.7 to 98.2]
  FHA [EU]/mL (n=239,240) | 96.7 [93.5 to 98.5] | 95.0 [91.4 to 97.4]
  PT [EU]/mL (n=239,240) | 94.1 [90.4 to 96.8] | 95.0 [91.4 to 97.4]
  PRN [EU]/mL (n=239,240) | 93.7 [89.9 to 96.4] | 95.8 [92.5 to 98.0]
Statistical Analysis 1: Comparison: 13vPnC vs 7vPnC; For Haemophilus influenzae type b the difference in percentage between the two groups (13vPnC - 7vPnC) at 0.15μg/mL threshold was calculated; Test type: Non-Inferiority or Equivalence — Non-inferiority for concomitant antigens was declared if the lowest limit of 2-sided 95% CI for the difference between the 2 groups (13vPnC - 7vPnC) was > -10%; Difference = 0.1, 95% CI [-2.9 to 3.1]
Statistical Analysis 2: Comparison: 13vPnC vs 7vPnC; For Haemophilus influenzae type b the difference in percentage between the two groups (13vPnC - 7vPnC) at 1.0 μg/mL threshold was calculated; Test type: Non-Inferiority or Equivalence — [test comment as in outcome 3, analysis 1]; Difference = -0.6, 95% CI [-8.3 to 7.0]
Statistical Analysis 3: Comparison: 13vPnC vs 7vPnC; For diphtheria toxoid the difference in percentage between the two groups (13vPnC - 7vPnC) at 0.1 IU/mL threshold was calculated; Test type: Non-Inferiority or Equivalence — [test comment as in outcome 3, analysis 1]; Difference = -0.4, 95% CI [-4.3 to 3.5]
Statistical Analysis 4: Comparison: 13vPnC vs 7vPnC; For Pertussis FHA the difference in percentage between the two groups (13vPnC - 7vPnC) at 40.5 EU/mL threshold was calculated; Test type: Non-Inferiority or Equivalence — [test comment as in outcome 3, analysis 1]; Difference = 1.7, 95% CI [-2.1 to 5.6]
Statistical Analysis 5: Comparison: 13vPnC vs 7vPnC; For Pertussis PT the difference in percentage between the two groups (13vPnC - 7vPnC) at 16.5 EU/mL threshold was calculated; Test type: Non-Inferiority or Equivalence — [test comment as in outcome 3, analysis 1]; Difference = -0.9, 95% CI [-5.2 to 3.4]
Statistical Analysis 6: Comparison: 13vPnC vs 7vPnC; For Pertussis PRN the difference in percentage between the two groups (13vPnC - 7vPnC) at 26 EU/mL threshold was calculated; Test type: Non-Inferiority or Equivalence — [test comment as in outcome 3, analysis 1]; Difference = -2.1, 95% CI [-6.4 to 2.0]

4. Secondary Outcome: Percentage of Participants Achieving Predefined Antibody Levels for Concomitant Vaccine Antigens Induced by Measles, Mumps, Rubella, Varicella (MMR-V) and Haemophilus Influenzae Type b (Hib)
Time Frame: One month after toddler dose (13 to 16 months of age)
Population: Evaluable immunogenicity (per protocol) population of eligible participants who adhered to the protocol requirements, had valid and determinate assay results, and had no other major protocol violations.(n)=number of participants with a determinate posttoddler dose antibody concentration to the given concomitant antigen.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | 13vPnC | 7vPnC
Number analyzed (Participants) | 239 | 223
percentage of participants
  Measles ≥1.10 I.V. (n=221,210) | 96.4 [93.0 to 98.4] | 97.1 [93.9 to 98.9]
  Mumps ≥1.10 I.V. (n=221,210) | 76.5 [70.3 to 81.9] | 72.9 [66.3 to 78.7]
  Rubella ≥15 IU/mL (n=209,204) | 91.9 [87.3 to 95.2] | 90.7 [85.8 to 94.3]
  Varicella ≥1.09 I.V. (n=221,210) | 26.7 [21.0 to 33.0] | 21.9 [16.5 to 28.1]
  Hib (PRP) 0.15 µg/mL (n=230,214) | 100.0 [98.4 to 100.0] | 100.0 [98.3 to 100.0]
  Hib (PRP) 1.0 µg/mL (n=230,214) | 90.4 [85.9 to 93.9] | 92.1 [87.6 to 95.3]
Statistical Analysis 1: Comparison: 13vPnC vs 7vPnC; [analysis description as in outcome 3, analysis 1]; Test type: Non-Inferiority or Equivalence — Non-inferiority for concomitant antigens was declared if the lowest limit of 2-sided 95% CI for the difference between the 2 groups (13vPnC - 7vPnC) > -10%; Difference = 0.0, 95% CI [-1.6 to 1.7]
Statistical Analysis 2: Comparison: 13vPnC vs 7vPnC; For Haemophilus influenzae type b the difference in percentage between the two groups (13vPnC - 7vPnC) at 1.0μg/mL threshold was calculated; Test type: Non-Inferiority or Equivalence — [test comment as in outcome 4, analysis 1]; Difference = -1.6, 95% CI [-7.1 to 3.8]
Statistical Analysis 3: Comparison: 13vPnC vs 7vPnC; For Measles the difference in percentage between the two groups (13vPnC - 7vPnC) at ≥1.10 I.V. threshold was calculated; Test type: Non-Inferiority or Equivalence — Non-inferiority for concomitant antigens was declared if the lowest limit of 2-sided 95% CI for the difference between the 2 groups (13vPnC - 7vPnC) > -5%; Difference = -0.8, 95% CI [-4.5 to 2.9]
Statistical Analysis 4: Comparison: 13vPnC vs 7vPnC; For Mumps the difference in percentage between the two groups (13vPnC - 7vPnC) at ≥1.10 I.V. threshold was calculated; Test type: Non-Inferiority or Equivalence — [test comment as in outcome 4, analysis 3]; Difference = 3.6, 95% CI [-4.7 to 11.9]
Statistical Analysis 5: Comparison: 13vPnC vs 7vPnC; For Rubella the difference in percentage between the two groups (13vPnC - 7vPnC) at ≥15 IU/mL threshold was calculated; Test type: Non-Inferiority or Equivalence — [test comment as in outcome 4, analysis 3]; Difference = 1.2, 95% CI [-4.4 to 6.9]
Statistical Analysis 6: Comparison: 13vPnC vs 7vPnC; For Varicella the difference in percentage between the two groups (13vPnC - 7vPnC) at ≥1.09 I.V. threshold was calculated; Test type: Non-Inferiority or Equivalence — [test comment as in outcome 4, analysis 1]; Difference = 4.8, 95% CI [-3.4 to 13.0]

5. Secondary Outcome: Geometric Mean Antibody Concentration of Hib PRP in 13vPnC Group Relative to 7vPnC Group After the Toddler Dose
Time Frame: one month after the toddler dose
Population: The all-available toddler immunogenicity population included all subjects who had at least 1 valid and determinate assay result before (excluding postinfant) or after the toddler dose. N = number of participants with a determinate antibody concentration or index value for the specified concomitant antigen.
Measure: Geometric Mean (95% Confidence Interval); unit: µg/mL
Arm/Group | 13vPnC | 7vPnC
Number analyzed (Participants) | 248 | 231
µg/mL | 6.84 [5.85 to 7.99] | 7.30 [6.21 to 8.59]
Statistical Analysis 1: Comparison: 13vPnC vs 7vPnC; For Haemophilus influenzae type b (PRP) the GMC ratio (13vPnC/7vPnC) was calculated; Test type: Non-Inferiority or Equivalence — Non-inferiority for concomitant antigens was declared if the lower bound of the 2-sided, 95% CI for the GMC ratio (13vPnC group/7vPnC group) was >0.5 (2-fold criterion); Ratio = 0.94, 95% CI [0.75 to 1.17]

6. Secondary Outcome: Geometric Mean Antibody Concentration of Measles, Mumps, and Varicella ELISA in 13vPnC Group Relative to 7vPnC Group After the Toddler Dose
Description: Normalization was performed for unit of measure "index value" as Index Value of 1.00 = 10 mIU/mL.
Time Frame: one month after the toddler dose
Population: as for outcome 5
Measure: Geometric Mean (95% Confidence Interval); unit: index value
Arm/Group | 13vPnC | 7vPnC
Number analyzed (Participants) | 239 | 227
index value
  Measles | 1.98 [1.81 to 2.16] | 2.06 [1.90 to 2.23]
  Mumps | 1.32 [1.19 to 1.46] | 1.32 [1.20 to 1.45]
  Varicella | 0.74 [0.69 to 0.79] | 0.73 [0.69 to 0.77]
Statistical Analysis 1: Comparison: 13vPnC vs 7vPnC; For Measles the GMC ratio (13vPnC/7vPnC) was calculated; Test type: Non-Inferiority or Equivalence — [test comment as in outcome 5, analysis 1]; Ratio = 0.96, 95% CI 2-sided [0.85 to 1.08]
Statistical Analysis 2: Comparison: 13vPnC vs 7vPnC; For Mumps the GMC ratio (13vPnC/7vPnC) was calculated; Test type: Non-Inferiority or Equivalence — [test comment as in outcome 5, analysis 1]; Ratio = 1.00, 95% CI 2-sided [0.87 to 1.14]
Statistical Analysis 3: Comparison: 13vPnC vs 7vPnC; For Varicella the GMC ratio (13vPnC/7vPnC) was calculated; Test type: Non-Inferiority or Equivalence — [test comment as in outcome 5, analysis 1]; Ratio = 1.01, 95% CI 2-sided [0.92 to 1.10]

7. Secondary Outcome: Geometric Mean Antibody Concentration of Rubella in 13vPnC Group Relative to 7vPnC Group After the Toddler Dose
Time Frame: one month after the toddler dose
Population: as for outcome 5
Measure: Geometric Mean (95% Confidence Interval); unit: IU/mL
Arm/Group | 13vPnC | 7vPnC
Number analyzed (Participants) | 227 | 221
IU/mL | 76.53 [64.55 to 90.72] | 97.69 [82.28 to 115.98]
Statistical Analysis 1: Comparison: 13vPnC vs 7vPnC; For Rubella the GMC ratio (13vPnC/7vPnC) was calculated; Test type: Non-Inferiority or Equivalence — [test comment as in outcome 5, analysis 1]; Ratio = 0.78, 95% CI 2-sided [0.62 to 1.00]

8. Primary Outcome: Percentage of Participants Reporting Pre-specified Systemic Events
Description: Systemic events (any fever [Fv] ≥ 38 degrees Celsius [C], decreased (decr.) appetite, irritability, increased (incr.) sleep, decreased sleep, and hives [urticaria], use of antipyretic medication [med] to treat or prevent symptoms [sx]) were reported using an electronic diary. Participants may be represented in more than 1 category.
Time Frame: Within 7 days after each dose
Population: Safety population who received the given vaccination. (n)= number of participants reporting yes for at least 1 day or no for all days.
Measure: Number; unit: Percentage of participants
Groups:
- 13vPnC Dose 1: Participants received one single 0.5 mL dose of 13-valent pneumococcal conjugate vaccine (13vPnC) coadministered with Haemophilus b Conjugate Vaccine (ActHIB) and Diphtheria and Tetanus Toxoids and Acellular Pertussis Adsorbed, Hepatitis B (Recombinant) and Inactivated Poliovirus Vaccine Combined (Pediarix) at 2 months (infant series).
- 7vPnC Dose 1: Participants received one single 0.5 mL dose of 7-valent pneumococcal conjugate vaccine (7vPnC) coadministered with Haemophilus b Conjugate Vaccine (ActHIB) and Diphtheria and Tetanus Toxoids and Acellular Pertussis Adsorbed, Hepatitis B (Recombinant) and Inactivated Poliovirus Vaccine Combined (Pediarix) at 2 months (infant series).
- 13vPnC Dose 2: Participants received one single 0.5 mL dose of 13-valent pneumococcal conjugate vaccine (13vPnC) coadministered with Haemophilus b Conjugate Vaccine (ActHIB) and Diphtheria and Tetanus Toxoids and Acellular Pertussis Adsorbed, Hepatitis B (Recombinant) and Inactivated Poliovirus Vaccine Combined (Pediarix) at 4 months (infant series).
- 7vPnC Dose 2: Participants received one single 0.5 mL dose of 7-valent pneumococcal conjugate vaccine (7vPnC) coadministered with Haemophilus b Conjugate Vaccine (ActHIB) and Diphtheria and Tetanus Toxoids and Acellular Pertussis Adsorbed, Hepatitis B (Recombinant) and Inactivated Poliovirus Vaccine Combined (Pediarix) at 4 months (infant series).
- 13vPnC Dose 3: Participants received one single 0.5 mL dose of 13-valent pneumococcal conjugate vaccine (13vPnC) coadministered with Haemophilus b Conjugate Vaccine (ActHIB) and Diphtheria and Tetanus Toxoids and Acellular Pertussis Adsorbed, Hepatitis B (Recombinant) and Inactivated Poliovirus Vaccine Combined (Pediarix) at 6 months (infant series).
- 7vPnC Dose 3: Participants received one single 0.5 mL dose of 7-valent pneumococcal conjugate vaccine (7vPnC) coadministered with Haemophilus b Conjugate Vaccine (ActHIB) and Diphtheria and Tetanus Toxoids and Acellular Pertussis Adsorbed, Hepatitis B (Recombinant) and Inactivated Poliovirus Vaccine Combined (Pediarix) at 6 months (infant series).
- 13vPnC Toddler Dose: Participants received one single 0.5 mL dose of 13vPnC coadministered with measles, mumps, rubella varicella vaccine live (ProQuad), Haemophilus b Conjugate Vaccine (Meningococcal Protein Conjugate) (PedvaxHIB), and Hepatitis A Vaccine, Inactivated (VAQTA) at 12-15 months of age (toddler dose).
- 7vPnC Toddler Dose: Participants received one single 0.5 mL dose of 7vPnC coadministered with measles, mumps, rubella varicella vaccine live (ProQuad), Haemophilus b Conjugate Vaccine (Meningococcal Protein Conjugate) (PedvaxHIB), and Hepatitis A Vaccine, Inactivated (VAQTA) at 12-15 months of age (toddler dose).
Arm/Group | 13vPnC Dose 1 | 7vPnC Dose 1 | 13vPnC Dose 2 | 7vPnC Dose 2 | 13vPnC Dose 3 | 7vPnC Dose 3 | 13vPnC Toddler Dose | 7vPnC Toddler Dose
Number analyzed (Participants) | 332 | 331 | 309 | 305 | 298 | 300 | 272 | 265
Percentage of participants
  Fv≥38°C but ≤39°C(n=196,203,146,151,123,106,99,76 | 24.0 | 21.2 | 43.2 | 40.4 | 39.8 | 37.7 | 53.5 | 51.3
  Fv>39°C but ≤40°C(n=177,187,118,123,94,81,61,48) | 2.8 | 0.0 | 2.5 | 4.9 | 8.5 | 2.5 | 6.6 | 12.5
  Fv >40°C (n=174,187,116,121,87,80,60,45) | 0.0 | 0.0 | 0.0 | 0.8 | 0.0 | 1.3 | 1.7 | 0.0
  Decr. appetite (n=228,238,177,174,147,136,116,110) | 54.8 | 45.4 | 59.9 | 52.3 | 59.2 | 59.6 | 65.5 | 73.6
  Irritability (n=289,290,236,236,216,218,199,175) | 89.6 | 85.9 | 89.8 | 91.5 | 88.4 | 92.2 | 92.0 | 93.1
  Incr. sleep (n=268,270,203,200,164,149,115,109) | 79.5 | 78.5 | 79.3 | 73.5 | 71.3 | 69.8 | 70.4 | 74.3
  Decr. sleep (n=221,236,169,172,154,134,113,95) | 45.7 | 47.9 | 49.1 | 55.8 | 60.4 | 63.4 | 58.4 | 64.2
  Hives (urticaria) (n=178,188,118,120,89,79,62,47) | 1.7 | 1.1 | 2.5 | 0.0 | 4.5 | 0.0 | 4.8 | 6.4
  Med-treat sx (n=257,266,221,221,203,187,162,138) | 78.6 | 71.8 | 82.4 | 81.9 | 82.3 | 85.6 | 84.0 | 87.7
  Med-prevent sx (n=272,274,233,231,202,189,164,162) | 75.0 | 74.8 | 86.7 | 83.5 | 81.2 | 84.1 | 88.4 | 90.7

9. Primary Outcome: Percentage of Participants Reporting Pre-specified Local Reactions
Description: Local reactions were reported using an electronic diary. Tenderness was scaled as Any (tenderness present); Significant ([Sig.], present and interfered with limb movement). Redness and swelling were scaled as Any (redness or swelling present); Mild (0.5 centimeters [cm] to 2.0 cm); Moderate ([Mod.], 2.5 to 7.0 cm); Severe ([Sev.], > 7.0 cm). Participants may have been represented in more than 1 category.
Time Frame: Within 7 days after each dose
Population: as for outcome 8
Measure: Number; unit: Percentage of participants
Groups:
- 7vPnC Toddler Series: Participants received one single 0.5 mL dose of 7vPnC coadministered with measles, mumps, rubella varicella vaccine live (ProQuad), Haemophilus b Conjugate Vaccine (Meningococcal Protein Conjugate) (PedvaxHIB), and Hepatitis A Vaccine, Inactivated (VAQTA) at 12-15 months of age (toddler dose).
Arm/Group | 13vPnC Dose 1 | 7vPnC Dose 1 | 13vPnC Dose 2 | 7vPnC Dose 2 | 13vPnC Dose 3 | 7vPnC Dose 3 | 13vPnC Toddler Dose | 7vPnC Toddler Series
Number analyzed (Participants) | 332 | 331 | 309 | 305 | 298 | 300 | 272 | 265
Percentage of participants
  Tenderness-Any (n=264,270,200,216,178,173,149,147) | 72.7 | 72.2 | 77.0 | 75.9 | 78.7 | 80.9 | 81.2 | 84.4
  Tenderness-Sig. (n=182,195,123,131,91,86,65,49) | 13.7 | 9.2 | 10.6 | 11.5 | 8.8 | 9.3 | 15.4 | 12.2
  Swelling-Any (n=201,216,141,146,116,103,91,73) | 27.4 | 23.6 | 31.2 | 29.5 | 37.9 | 36.9 | 44.0 | 50.7
  Swelling-Mild (n=199,212,141,142,113,103,90,71) | 23.1 | 21.2 | 29.8 | 26.1 | 35.4 | 36.9 | 43.3 | 46.5
  Swelling-Mod. (n=176,193,118,126,91,82,68,49) | 6.8 | 5.2 | 5.1 | 7.1 | 6.6 | 6.1 | 14.7 | 14.3
  Swelling-Sev. (n=172,187,116,120,87,79,59,44) | 0.0 | 0.0 | 0.0 | 0.0 | 0.0 | 0.0 | 0.0 | 0.0
  Redness-Any (n=202,223,155,164,131,118,103,87) | 35.6 | 32.3 | 45.2 | 37.8 | 48.9 | 50.0 | 54.4 | 65.5
  Redness-Mild (n=200,220,155,162,128,117,102,85) | 34.5 | 31.4 | 44.5 | 37.0 | 47.7 | 48.7 | 53.9 | 63.5
  Redness-Mod. (n=177,191,117,124,91,80,62,50) | 4.5 | 2.6 | 1.7 | 3.2 | 5.5 | 5.0 | 8.1 | 14.0
  Redness-Sev. (n=173,186,116,120,87,79,59,44) | 0.0 | 0.0 | 0.0 | 0.0 | 0.0 | 0.0 | 0.0 | 0.0

10. Secondary Outcome: Percentage of Participants Achieving Functional Antibody Titer ≥1:8 as Measured by Opsonophagocytic Activity Assay (OPA) in 13vPnC Group Relative to 7vPnC Group the 3-Dose Infant Series and the Toddler Dose
Description: Percentage of participants achieving functional antibody titer ≥1:8 as measured by opsonophagocytic activity assay (OPA) along with the corresponding 95% CI for the 7 common pneumococcal serotypes (serotypes 4, 6B, 9V, 14, 18C, 19F, and 23F) and 6 additional pneumococcal serotypes specific to 13vPnC (serotypes 1, 3, 5, 6A, 7F, and 19A) are presented.
Time Frame: One month after infant series and one month after toddler dose
Population: Evaluable immunogenicity (per protocol) population of eligible participants who adhered to the protocol requirements, had valid and determinate assay results, and had no other major protocol violations;(n) = number of participants with a determinate postinfant series OPA antibody titer to the given serotype.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Groups:
- 13vPnC After Infant Series; 7vPnC After Infant Series; 13vPnC After Toddler Dose; 7vPnC After Toddler Dose: Participants received 1 single 0.5 mL dose together with a concomitant dose of Pediarix and ActHIB at the 2-, 4-, and 6-month visits and ProQuad, PedvaxHIB, and VAQTA at the 12-15 month visit.
Arm/Group | 13vPnC After Infant Series | 7vPnC After Infant Series | 13vPnC After Toddler Dose | 7vPnC After Toddler Dose
Number analyzed (Participants) | 252 | 252 | 239 | 223
percentage of participants
  Common Serotypes - Serotype 4 (n=92,92,88,92) | 97.8 [92.4 to 99.7] | 98.9 [94.1 to 100.0] | 98.9 [93.8 to 100.0] | 98.9 [94.1 to 100.0]
  Common Serotypes - Serotype 6B (n=94,94,92,95) | 98.9 [94.2 to 100.0] | 100.0 [96.2 to 100.0] | 98.9 [94.1 to 100.0] | 100.0 [96.2 to 100.0]
  Common Serotypes - Serotype 9V (n=93,94,90,94) | 100.0 [96.1 to 100.0] | 98.9 [94.2 to 100.0] | 98.9 [94.0 to 100.0] | 100.0 [96.2 to 100.0]
  Common Serotypes - Serotype 14 (n=94,94,92,96) | 100.0 [96.2 to 100.0] | 100.0 [96.2 to 100.0] | 100.0 [96.1 to 100.0] | 100.0 [96.2 to 100.0]
  Common Serotypes - Serotype 18C (n=94,94,91,96) | 100.0 [96.2 to 100.0] | 100.0 [96.2 to 100.0] | 98.9 [94.0 to 100.0] | 100.0 [96.2 to 100.0]
  Common Serotypes - Serotype 19F (n=94,94,92,96) | 90.4 [82.6 to 95.5] | 92.6 [85.3 to 97.0] | 96.7 [90.8 to 99.3] | 94.8 [88.3 to 98.3]
  Common Serotypes - Serotype 23F (n=94,94,90,92) | 98.9 [94.2 to 100.0] | 98.9 [94.2 to 100.0] | 98.9 [94.0 to 100.0] | 100.0 [96.1 to 100.0]
  Additional Serotypes - Serotype 1 (n=92,92,89,92) | 98.9 [94.1 to 100.0] | 9.8 [4.6 to 17.8] | 98.9 [93.9 to 100.0] | 12.0 [6.1 to 20.4]
  Additional Serotypes - Serotype 3 (n=94,94,91,96) | 96.8 [91.0 to 99.3] | 21.3 [13.5 to 30.9] | 97.8 [92.3 to 99.7] | 43.8 [33.6 to 54.3]
  Additional Serotypes - Serotype 5 (n=91,93,91,96) | 92.3 [84.8 to 96.9] | 2.2 [0.3 to 7.6] | 98.9 [94.0 to 100.0] | 5.2 [1.7 to 11.7]
  Additional Serotypes - Serotype 6A (n=94,94,92,96) | 100.0 [96.2 to 100.0] | 77.7 [67.9 to 85.6] | 98.9 [94.1 to 100.0] | 94.8 [88.3 to 98.3]
  Additional Serotypes - Serotype 7F (n=94,89,91,92) | 100.0 [96.2 to 100.0] | 76.4 [66.2 to 84.8] | 100.0 [96.0 to 100.0] | 80.4 [70.9 to 88.0]
  Additional Serotypes-Serotype 19A (n=93,92,91,94) | 91.4 [83.8 to 96.2] | 16.3 [9.4 to 25.5] | 97.8 [92.3 to 99.7] | 53.2 [42.6 to 63.6]

11. Secondary Outcome: Geometric Mean Titer (GMT) as Measured by Opsonophagocytic Activity Assay (OPA) in 13vPnC Group Relative to 7vPnC Group After the 3-Dose Infant Series and the Toddler Dose
Description: Geometric mean titer (GMT) as measured by opsonophagocytic activity assay (OPA) for 7 common pneumococcal serotypes (serotypes 4, 6B, 9V, 14, 18C, 19F, and 23F) and 6 additional pneumococcal serotypes specific to 13vPnC (Serotypes 1, 3, 5, 6A, 7F, and 19A) are presented.
Time Frame: one month after the infant series and the toddler dose
Population: Evaluable immunogenicity (per protocol) population of eligible subjects who adhered to the protocol requirements, had valid and determinate assay results, and had no other major protocol violations, (n) = number of participants with a determinate antibody titer for the specified serotype.
Measure: Geometric Mean (95% Confidence Interval); unit: titer
Groups:
- 13vPnC After the Infant Series; 13vPnC After the Toddler Dose: Subjects received 1 single 0.5 mL dose of 13vPnC coadministered with Pediarix and ActHIB at the 2-, 4-, and 6-month visits and ProQuad, PedvaxHIB, and VAQTA at the 12-15 month visit.
- 7vPnC After the Infant Series; 7vPnC After the Toddler Dose: Subjects received 1 single 0.5 mL dose of 7vPnC coadministered with Pediarix and ActHIB at the 2-, 4-, and 6-month visits and ProQuad, PedvaxHIB, and VAQTA at the 12-15 month visit.
Arm/Group | 13vPnC After the Infant Series | 7vPnC After the Infant Series | 13vPnC After the Toddler Dose | 7vPnC After the Toddler Dose
Number analyzed (Participants) | 252 | 252 | 239 | 223
titer
  Common Serotypes -Serotype 4 (n=92,92,88,92) | 359.32 [276.04 to 467.72] | 535.68 [421.13 to 681.37] | 1179.98 [847.34 to 1643.20] | 1492.46 [1114.40 to 1998.78]
  Common Serotypes - Serotype 6B (n=94,94,92,95) | 1054.65 [817.34 to 1360.87] | 1513.66 [1206.64 to 1898.81] | 3099.51 [2337.02 to 4110.79] | 4066.22 [3243.42 to 5097.76]
  Common Serotypes - Serotype 9V (n=93,94,90,94) | 4035.40 [2932.68 to 5552.75] | 3259.01 [2288.43 to 4641.25] | 11856.03 [8809.85 to 15955.49] | 18032.33 [14124.99 to 23020.53]
  Common Serotypes - Serotype 14 (n=94,94,92,96) | 1240.41 [934.93 to 1645.69] | 1480.55 [1133.40 to 1934.02] | 2002.23 [1452.54 to 2759.93] | 2365.87 [1870.56 to 2992.34]
  Common Serotypes - Serotype 18C (n=94,94,91,96) | 275.59 [210.33 to 361.10] | 375.64 [291.68 to 483.75] | 993.27 [754.08 to 1308.33] | 1722.16 [1326.59 to 2235.67]
  Common Serotypes - Serotype 19F (n=94,94,92,96) | 54.42 [40.20 to 73.65] | 44.92 [33.90 to 59.52] | 199.65 [144.22 to 276.38] | 167.20 [121.35 to 230.37]
  Common Serotypes - Serotype 23F (n=94,94,90,92) | 791.07 [604.96 to 1034.44] | 923.56 [708.59 to 1203.74] | 2723.25 [1960.67 to 3782.41] | 4981.68 [3885.71 to 6386.76]
  Additional Serotypes - Serotype 1 (n=92,92,89,92) | 51.83 [38.84 to 69.16] | 4.41 [4.06 to 4.80] | 164.23 [113.83 to 236.93] | 5.01 [4.22 to 5.96]
  Additional Serotypes - Serotype 3 (n=94,94,91,96) | 120.67 [92.38 to 157.62] | 6.70 [5.27 to 8.52] | 380.41 [300.19 to 482.08] | 11.81 [8.68 to 16.08]
  Additional Serotypes - Serotype 5 (n=91,93,91,96) | 90.86 [67.10 to 123.02] | 4.15 [3.94 to 4.38] | 300.41 [229.39 to 393.40] | 4.69 [3.99 to 5.51]
  Additional Serotypes - Serotype 6A (n=94,94,92,96) | 979.68 [783.04 to 1225.71] | 100.35 [66.22 to 152.08] | 2241.79 [1706.71 to 2944.63] | 538.54 [374.83 to 773.75]
  Additional Serotypes - Serotype 7F (n=94,89,91,92) | 9493.77 [7339.13 to 12280.98] | 128.00 [79.55 to 205.97] | 11629.44 [9053.62 to 14938.11] | 267.84 [164.49 to 436.11]
  Additional Serotypes-Serotype 19A (n=93,92,91,94) | 151.94 [105.16 to 219.52] | 6.53 [5.01 to 8.50] | 1024.00 [774.12 to 1354.54] | 28.65 [18.58 to 44.17]

ADVERSE EVENTS:
Time Frame: Adverse events were collected throughout the study.
Groups:
- 13vPnC Infant Series: Participants received one single 0.5 mL dose of 13-valent pneumococcal conjugate vaccine (13vPnC) coadministered with Haemophilus b Conjugate Vaccine (ActHIB) and Diphtheria and Tetanus Toxoids and Acellular Pertussis Adsorbed, Hepatitis B (Recombinant) and Inactivated Poliovirus Vaccine Combined (Pediarix) at 2 months (infant series).
- 7vPnC Infant Series: Participants received one single 0.5 mL dose of 7-valent pneumococcal conjugate vaccine (7vPnC) coadministered with Haemophilus b Conjugate Vaccine (ActHIB) and Diphtheria and Tetanus Toxoids and Acellular Pertussis Adsorbed, Hepatitis B (Recombinant) and Inactivated Poliovirus Vaccine Combined (Pediarix) at 2 months (infant series).
- 13vPnC Post Infant Series; 7vPnC Post Infant Series; 13vPnC 6-Month Follow-up; 7vPnC 6-Month Follow-up: Participants received 1 single 0.5 mL dose together with a concomitant dose of Pediarix and ActHIB at the 2-, 4-, and 6-month visits and ProQuad, PedvaxHIB, and VAQTA at the 12-15 month visit.
- 13vPnC Toddler Series: Participants received one single 0.5 mL dose of 13vPnC coadministered with measles, mumps, rubella varicella vaccine live (ProQuad), Haemophilus b Conjugate Vaccine (Meningococcal Protein Conjugate) (PedvaxHIB), and Hepatitis A Vaccine, Inactivated (VAQTA) at 12-15 months of age (toddler dose).
Arm/Group | 13vPnC Infant Series | 7vPnC Infant Series | 13vPnC Post Infant Series | 7vPnC Post Infant Series | 13vPnC Toddler Series | 7vPnC Toddler Series | 13vPnC 6-Month Follow-up | 7vPnC 6-Month Follow-up
Serious Adverse Events (participants affected / at risk) | 17/332 | 16/331 | 5/332 | 7/330 | 3/267 | 4/258 | 9/330 | 5/329
Other Adverse Events (participants affected / at risk) | 272/332 | 263/331 | 31/332 | 29/330 | 183/267 | 163/258 | 11/330 | 10/329
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | 13vPnC Infant Series (N=332) | 7vPnC Infant Series (N=331) | 13vPnC Post Infant Series (N=332) | 7vPnC Post Infant Series (N=330) | 13vPnC Toddler Series (N=267) | 7vPnC Toddler Series (N=258) | 13vPnC 6-Month Follow-up (N=330) | 7vPnC 6-Month Follow-up (N=329)
Abscess neck (Infections and infestations) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Accidental exposure (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Accidental overdose (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Apnoea (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Asthma (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 1
Bronchial hyperreactivity (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Bronchiolitis (Infections and infestations) | 4 | 6 | 0 | 2 | 0 | 0 | 1 | 0
Bronchitis (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Cellulitis (Infections and infestations) | 0 | 0 | 1 | 0 | 0 | 0 | 1 | 0
Congenital megacolon (Congenital, familial and genetic disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Constipation (Gastrointestinal disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Contusion (Injury, poisoning and procedural complications) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Convulsion (Nervous system disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Cough (Respiratory, thoracic and mediastinal disorders) | 1 | 1 | 0 | 0 | 0 | 1 | 0 | 0
Croup infectious (Infections and infestations) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Dehydration (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Epilepsy (Nervous system disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Febrile convulsion (Nervous system disorders) | 1 | 0 | 1 | 0 | 0 | 1 | 0 | 0
Femur fracture (Injury, poisoning and procedural complications) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Gastroenteritis (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Gastroenteritis viral (Infections and infestations) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Mastoiditis (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1
Nasopharyngitis (Infections and infestations) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Near drowning (Injury, poisoning and procedural complications) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Nephroblastoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Otitis media (Infections and infestations) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Pneumonia (Infections and infestations) | 1 | 0 | 0 | 1 | 0 | 0 | 1 | 0
Pneumonia respiratory syncytial viral (Infections and infestations) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Pneumonia viral (Infections and infestations) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Postical paralysis (Nervous system disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Pyrexia (General disorders) | 2 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Rectal abscess (Infections and infestations) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Respiratory distress (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Respiratory syncytial virus bronchiolitis (Infections and infestations) | 3 | 2 | 0 | 0 | 0 | 0 | 1 | 1
Respiratory syncytial virus infection (Infections and infestations) | 0 | 2 | 0 | 0 | 0 | 0 | 1 | 0
Rhinitis (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Selective IgA immunodeficiency (Immune system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Skull fracture (Injury, poisoning and procedural complications) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Status asthmaticus (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | 2 | 1 | 0 | 0 | 1
Subcutaneous abscess (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Thromboycytopenia (Blood and lymphatic system disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Tibia fracture (Injury, poisoning and procedural complications) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Urinary tract infection (Infections and infestations) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Varicella (Infections and infestations) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Vomiting (Gastrointestinal disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk, or affected / at risk where a term's number at risk differs (number of events):
Term (organ system) | 13vPnC Infant Series (N=332) | 7vPnC Infant Series (N=331) | 13vPnC Post Infant Series (N=332) | 7vPnC Post Infant Series (N=330) | 13vPnC Toddler Series (N=267) | 7vPnC Toddler Series (N=258) | 13vPnC 6-Month Follow-up (N=330) | 7vPnC 6-Month Follow-up (N=329)
Anaemia (Blood and lymphatic system disorders) | 2 | 0 | 0 | 0 | 2 | 1 | 1 | 0
Lymphadenopathy (Blood and lymphatic system disorders) | 0 | 2 | 0 | 0 | 0 | 0 | 0 | 0
Neutropenia (Blood and lymphatic system disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Iron deficiency anaemia (Blood and lymphatic system disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Neutrophilia (Blood and lymphatic system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Plagiocephaly (Congenital, familial and genetic disorders) | 3 | 6 | 1 | 0 | 0 | 0 | 0 | 0
Ankyloglossia congenital (Congenital, familial and genetic disorders) | 1 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Macrocephaly (Congenital, familial and genetic disorders) | 1 | 1 | 0 | 0 | 0 | 0 | 2 | 1
Dermoid cyst (Congenital, familial and genetic disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Hydrocele (Congenital, familial and genetic disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Patent ductus arteriosus (Congenital, familial and genetic disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Pectus excavatum (Congenital, familial and genetic disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Phimosis (Congenital, familial and genetic disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Pilonidal cyst congenital (Congenital, familial and genetic disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Thalassaemia trait (Congenital, familial and genetic disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Atrial septal defect (Congenital, familial and genetic disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Hip dysplasia (Congenital, familial and genetic disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Sickle cell trait (Congenital, familial and genetic disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Haemoglobin C trait (Congenital, familial and genetic disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Talipes (Congenital, familial and genetic disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Tibial torsion (Congenital, familial and genetic disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Ear pain (Ear and labyrinth disorders) | 5 | 6 | 0 | 0 | 1 | 2 | 0 | 0
Cerumen impaction (Ear and labyrinth disorders) | 4 | 4 | 0 | 0 | 0 | 1 | 0 | 0
Middle ear effusion (Ear and labyrinth disorders) | 3 | 1 | 0 | 0 | 0 | 0 | 1 | 0
Eustachian tube dysfunction (Ear and labyrinth disorders) | 0 | 2 | 0 | 0 | 0 | 0 | 0 | 0
Tympanic membrane perforation (Ear and labyrinth disorders) | 1 | 1 | 0 | 0 | 0 | 1 | 0 | 0
Precocious puberty (Endocrine disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Conjunctivitis (Eye disorders) | 22 | 24 | 1 | 0 | 3 | 6 | 0 | 0
Eye discharge (Eye disorders) | 4 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Eye swelling (Eye disorders) | 3 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Strabismus (Eye disorders) | 2 | 1 | 1 | 0 | 0 | 0 | 0 | 0
Lacrimation increased (Eye disorders) | 0 | 2 | 0 | 0 | 0 | 0 | 0 | 0
Dacryostenosis acquired (Eye disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Eyelid irritation (Eye disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Scleral haemorrhage (Eye disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Diarrhoea (Gastrointestinal disorders) | 35 | 31 | 2 | 0 | 9 | 8 | 0 | 0
Vomiting (Gastrointestinal disorders) | 23 | 25 | 0 | 0 | 3 | 6 | 0 | 0
Constipation (Gastrointestinal disorders) | 16 | 21 | 0 | 0 | 2 | 1 | 0 | 0
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 11 | 23 | 1 | 0 | 0 | 0 | 0 | 0
Teething (Gastrointestinal disorders) | 4 | 7 | 0 | 1 | 3 | 2 | 0 | 0
Flatulence (Gastrointestinal disorders) | 3 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Abdominal pain (Gastrointestinal disorders) | 1 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Abdominal pain upper (Gastrointestinal disorders) | 0 | 2 | 0 | 0 | 0 | 0 | 0 | 0
Anal fissure (Gastrointestinal disorders) | 1 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Infantile spitting up (Gastrointestinal disorders) | 0 | 2 | 0 | 0 | 0 | 0 | 0 | 0
Inguinal hernia (Gastrointestinal disorders) | 1 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Nausea (Gastrointestinal disorders) | 0 | 2 | 0 | 0 | 0 | 0 | 0 | 0
Umbilical hernia (Gastrointestinal disorders) | 1 | 1 | 1 | 0 | 0 | 0 | 0 | 0
Abdominal wall disorder (Gastrointestinal disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Dysphagia (Gastrointestinal disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Faeces discoloured (Gastrointestinal disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Gingival cyst (Gastrointestinal disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Rectal fissure (Gastrointestinal disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Stomach discomfort (Gastrointestinal disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Anal skin tags (Gastrointestinal disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Enamel anomaly (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Ileus (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Pyrexia (General disorders) | 29 | 21 | 1 | 1 | 10 | 10 | 0 | 0
Irritability (General disorders) | 4 | 7 | 0 | 0 | 1 | 1 | 0 | 0
Injection site erythema (General disorders) | 2 | 1 | 0 | 0 | 2 | 1 | 0 | 0
Injection site swelling (General disorders) | 2 | 1 | 0 | 0 | 2 | 1 | 0 | 0
Injection site bruising (General disorders) | 1 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Injection site induration (General disorders) | 1 | 1 | 0 | 0 | 0 | 1 | 0 | 0
Xerosis (General disorders) | 1 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Developmental delay (General disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Hernia (General disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Influenza like illness (General disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Injection site pain (General disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Injection site rash (General disorders) | 0 | 1 | 0 | 0 | 1 | 0 | 0 | 0
Injection site reaction (General disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Oedema peripheral (General disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Allergy to metals (Immune system disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Drug hypersensitivity (Immune system disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Food allergy (Immune system disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 1
Hypersensitivity (Immune system disorders) | 0 | 1 | 1 | 0 | 0 | 1 | 0 | 0
Milk allergy (Immune system disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Seasonal allergy (Immune system disorders) | 1 | 0 | 1 | 1 | 0 | 0 | 0 | 0
Upper respiratory tract infection (Infections and infestations) | 131 | 131 | 3 | 2 | 21 | 24 | 1 | 0
Otitis media (Infections and infestations) | 94 | 77 | 3 | 4 | 23 | 23 | 1 | 0
Bronchiolitis (Infections and infestations) | 52 | 49 | 1 | 1 | 1 | 4 | 0 | 0
Nasopharyngitis (Infections and infestations) | 21 | 18 | 1 | 2 | 0 | 0 | 0 | 0
Viral upper respiratory tract infection (Infections and infestations) | 18 | 20 | 0 | 0 | 1 | 3 | 0 | 0
Otitis media acute (Infections and infestations) | 12 | 22 | 0 | 1 | 5 | 3 | 0 | 0
Viral infection (Infections and infestations) | 13 | 18 | 0 | 1 | 5 | 2 | 0 | 0
Candidiasis (Infections and infestations) | 11 | 16 | 0 | 0 | 0 | 1 | 0 | 0
Gastroenteritis (Infections and infestations) | 10 | 11 | 1 | 1 | 2 | 3 | 0 | 0
Sinusitis (Infections and infestations) | 12 | 6 | 0 | 0 | 1 | 3 | 0 | 0
Oral candidiasis (Infections and infestations) | 10 | 4 | 0 | 0 | 1 | 0 | 0 | 0
Pharyngitis (Infections and infestations) | 7 | 6 | 0 | 0 | 6 | 4 | 0 | 0
Rhinitis (Infections and infestations) | 5 | 8 | 1 | 0 | 1 | 1 | 0 | 0
Candida nappy rash (Infections and infestations) | 7 | 5 | 0 | 0 | 2 | 1 | 0 | 0
Pneumonia (Infections and infestations) | 7 | 5 | 0 | 0 | 2 | 1 | 1 | 0
Croup infectious (Infections and infestations) | 5 | 5 | 0 | 0 | 7 | 6 | 0 | 0
Respiratory syncytial virus infection (Infections and infestations) | 5 | 5 | 0 | 0 | 0 | 0 | 0 | 0
Viral skin infection (Infections and infestations) | 4 | 5 | 0 | 1 | 0 | 2 | 0 | 0
Gastroenteritis viral (Infections and infestations) | 4 | 4 | 0 | 0 | 1 | 0 | 0 | 0
Respiratory syncytial virus bronchiolitis (Infections and infestations) | 4 | 4 | 0 | 0 | 0 | 0 | 0 | 0
Bronchitis (Infections and infestations) | 4 | 2 | 0 | 0 | 0 | 2 | 0 | 0
Gastroenteritis rotavirus (Infections and infestations) | 4 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Skin candida (Infections and infestations) | 4 | 1 | 0 | 0 | 0 | 2 | 0 | 0
Conjunctivitis bacterial (Infections and infestations) | 1 | 3 | 0 | 0 | 0 | 1 | 0 | 0
Ear infection (Infections and infestations) | 3 | 1 | 0 | 0 | 0 | 2 | 0 | 0
Impetigo (Infections and infestations) | 3 | 1 | 1 | 0 | 1 | 0 | 0 | 0
Viral pharyngitis (Infections and infestations) | 2 | 2 | 1 | 0 | 0 | 0 | 0 | 0
Body tinea (Infections and infestations) | 2 | 1 | 0 | 1 | 2 | 0 | 0 | 0
Fungal skin infection (Infections and infestations) | 3 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Influenza (Infections and infestations) | 2 | 1 | 0 | 0 | 1 | 0 | 0 | 0
Intertrigo candida (Infections and infestations) | 2 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Tinea capitis (Infections and infestations) | 1 | 2 | 0 | 0 | 0 | 0 | 0 | 0
Urinary tract infection (Infections and infestations) | 0 | 3 | 0 | 0 | 0 | 0 | 0 | 0
Bronchiectasis (Infections and infestations) | 1 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Conjunctivitis viral (Infections and infestations) | 0 | 2 | 0 | 0 | 0 | 0 | 0 | 0
Ear lobe infection (Infections and infestations) | 2 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Eye infection (Infections and infestations) | 0 | 2 | 0 | 0 | 0 | 0 | 0 | 0
Folliculitis (Infections and infestations) | 2 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Genital candidiasis (Infections and infestations) | 1 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Pharyngitis streptococcal (Infections and infestations) | 0 | 2 | 0 | 0 | 0 | 1 | 0 | 0
Respiratory tract infection viral (Infections and infestations) | 2 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Acute sinusitis (Infections and infestations) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Breast cellulitis (Infections and infestations) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Bronchitis viral (Infections and infestations) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Conjunctivitis infective (Infections and infestations) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Eczema infected (Infections and infestations) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Enteritis infectious (Infections and infestations) | 0 | 1 | 0 | 0 | 0 | 1 | 0 | 0
Enterobiasis (Infections and infestations) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Erythema infectiosum (Infections and infestations) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Fungal infection (Infections and infestations) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Gastritis viral (Infections and infestations) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Laryngitis (Infections and infestations) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Otitis externa (Infections and infestations) | 0 | 1 | 0 | 0 | 2 | 0 | 0 | 0
Parainfluenzae virus infection (Infections and infestations) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Paronychia (Infections and infestations) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Rash pustular (Infections and infestations) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Roseola (Infections and infestations) | 1 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Staphylococcal infection (Infections and infestations) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Viraemia (Infections and infestations) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Otitis media chronic (Infections and infestations) | 0 | 0 | 1 | 1 | 0 | 0 | 0 | 0
Infected insect bite (Infections and infestations) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Tinea infection (Infections and infestations) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Varicella (Infections and infestations) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Wound infection staphylococcal (Infections and infestations) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
External ear cellulitis (Infections and infestations) | 0 | 0 | 0 | 0 | 2 | 0 | 0 | 0
Cellulitis (Infections and infestations) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Hand-foot-and-mouth disease (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Lice infestation (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Oral fungal infection (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Oral herpes (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Viral diarrhoea (Infections and infestations) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Rotavirus infection (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Contusion (Injury, poisoning and procedural complications) | 1 | 1 | 0 | 0 | 1 | 1 | 0 | 0
Fall (Injury, poisoning and procedural complications) | 1 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Thermal burn (Injury, poisoning and procedural complications) | 2 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Arthropod bite (Injury, poisoning and procedural complications) | 1 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Burns first degree (Injury, poisoning and procedural complications) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Excoriation (Injury, poisoning and procedural complications) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Injury (Injury, poisoning and procedural complications) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Lower limb fracture (Injury, poisoning and procedural complications) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Procedural pain (Injury, poisoning and procedural complications) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Road traffic accident (Injury, poisoning and procedural complications) | 1 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Skin laceration (Injury, poisoning and procedural complications) | 1 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Head injury (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 2 | 1 | 0 | 0
Animal bite (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Arthropod sting (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Cardiac murmur (Investigations) | 2 | 2 | 1 | 2 | 0 | 0 | 0 | 0
Blood thyroid stimulating hormone decreased (Investigations) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Cardiac murmur functional (Investigations) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Head circumference abnormal (Investigations) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Weight decreased (Investigations) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Dehydration (Metabolism and nutrition disorders) | 1 | 3 | 0 | 0 | 1 | 2 | 0 | 0
Food intolerance (Metabolism and nutrition disorders) | 2 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Anorexia (Metabolism and nutrition disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Decreased appetite (Metabolism and nutrition disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Failure to thrive (Metabolism and nutrition disorders) | 1 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Obesity (Metabolism and nutrition disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Weight gain poor (Metabolism and nutrition disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Lactose intolerance (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Torticollis (Musculoskeletal and connective tissue disorders) | 2 | 2 | 0 | 0 | 0 | 0 | 0 | 0
Muscular weakness (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Nose deformity (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Weight bearing difficulty (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Premature closure of cranial sutures (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Haemangioma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Melanocytic naevus (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 2 | 0 | 0 | 0 | 0 | 0 | 0
Benign vaginal neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Haemangioma of skin (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Skin papilloma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Tremor (Nervous system disorders) | 1 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Convulsion (Nervous system disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Headache (Nervous system disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Hypersomnia (Nervous system disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Hypertonia (Nervous system disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Hypokinesia (Nervous system disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Lethargy (Nervous system disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Nystagmus (Nervous system disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Somnolence (Nervous system disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Speech disorder developmental (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Crying (Psychiatric disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Insomnia (Psychiatric disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Restlessness (Psychiatric disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Staring (Psychiatric disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Crystalluria (Renal and urinary disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Vesicoureteric reflux (Renal and urinary disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Penile adhesion (Reproductive system and breast disorders) | 3 | 2 | 0 | 0 | 1 | 0 | 0 | 0
Vulval disorder (Reproductive system and breast disorders) | 1 | 3 | 0 | 0 | 0 | 0 | 0 | 0
Genital discomfort (Reproductive system and breast disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Genital erythema (Reproductive system and breast disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Gynaecomastia (Reproductive system and breast disorders) | 1 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Penile blister (Reproductive system and breast disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Penis disorder (Reproductive system and breast disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Testicular retraction (Reproductive system and breast disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Cough (Respiratory, thoracic and mediastinal disorders) | 28 | 39 | 0 | 0 | 9 | 9 | 0 | 0
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 36 | 25 | 0 | 0 | 2 | 3 | 0 | 0
Rhinorrhoea (Respiratory, thoracic and mediastinal disorders) | 16 | 17 | 1 | 1 | 5 | 4 | 0 | 0
Wheezing (Respiratory, thoracic and mediastinal disorders) | 11 | 14 | 0 | 0 | 1 | 3 | 0 | 0
Bronchial hyperreactivity (Respiratory, thoracic and mediastinal disorders) | 6 | 9 | 0 | 0 | 0 | 3 | 0 | 0
Rhinitis allergic (Respiratory, thoracic and mediastinal disorders) | 4 | 6 | 1 | 3 | 3 | 2 | 1 | 0
Sinus congestion (Respiratory, thoracic and mediastinal disorders) | 2 | 4 | 1 | 0 | 0 | 0 | 0 | 0
Asthma (Respiratory, thoracic and mediastinal disorders) | 1 | 4 | 3 | 3 | 0 | 1 | 2 | 4
Choking (Respiratory, thoracic and mediastinal disorders) | 1 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 1 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Upper respiratory tract congestion (Respiratory, thoracic and mediastinal disorders) | 0 | 2 | 0 | 0 | 0 | 0 | 0 | 0
Apnoea (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Bronchospasm (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Dysphonia (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Haemoptysis (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Laryngospasm (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Lung infiltration (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Postnasal drip (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Respiratory distress (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Sleep apnoea syndrome (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Tachypnoea (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Pharyngolaryngeal pain (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Eczema (Skin and subcutaneous tissue disorders) | 31 | 31 | 1 | 4 | 1 | 3 | 1 | 2
Dermatitis diaper (Skin and subcutaneous tissue disorders) | 21 | 13 | 2 | 0 | 6 | 6 | 0 | 0
Seborrhoeic dermatitis (Skin and subcutaneous tissue disorders) | 7 | 17 | 1 | 0 | 0 | 0 | 0 | 0
Rash (Skin and subcutaneous tissue disorders) | 8 | 13 | 0 | 1 | 3 | 9 | 0 | 0
Dermatitis atopic (Skin and subcutaneous tissue disorders) | 7 | 12 | 0 | 0 | 1 | 0 | 1 | 0
Dry skin (Skin and subcutaneous tissue disorders) | 6 | 7 | 0 | 0 | 0 | 1 | 0 | 0
Seborrhoea (Skin and subcutaneous tissue disorders) | 3 | 5 | 0 | 0 | 0 | 0 | 0 | 0
Dermatitis (Skin and subcutaneous tissue disorders) | 3 | 3 | 1 | 0 | 1 | 0 | 0 | 0
Rash papular (Skin and subcutaneous tissue disorders) | 0 | 3 | 0 | 0 | 1 | 0 | 0 | 0
Acne infantile (Skin and subcutaneous tissue disorders) | 1 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Dandruff (Skin and subcutaneous tissue disorders) | 0 | 2 | 0 | 0 | 0 | 0 | 0 | 0
Dermatitis contact (Skin and subcutaneous tissue disorders) | 2 | 0 | 0 | 0 | 2 | 2 | 0 | 0
Drug eruption (Skin and subcutaneous tissue disorders) | 1 | 1 | 0 | 0 | 1 | 0 | 0 | 0
Rash erythematous (Skin and subcutaneous tissue disorders) | 1 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Urticaria (Skin and subcutaneous tissue disorders) | 0 | 2 | 0 | 0 | 0 | 1 | 0 | 0
Blister (Skin and subcutaneous tissue disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Cafe au lait spots (Skin and subcutaneous tissue disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Dermatitis allergic (Skin and subcutaneous tissue disorders) | 1 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Erythema (Skin and subcutaneous tissue disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Hyperhidrosis (Skin and subcutaneous tissue disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Intertrigo (Skin and subcutaneous tissue disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Pityriasis alba (Skin and subcutaneous tissue disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Post inflammatory pigmentation change (Skin and subcutaneous tissue disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Skin disorder (Skin and subcutaneous tissue disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Skin exfoliation (Skin and subcutaneous tissue disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Skin hyperpigmentation (Skin and subcutaneous tissue disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Skin hypopigmentation (Skin and subcutaneous tissue disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Skin lesion (Skin and subcutaneous tissue disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Umbilical erythema (Skin and subcutaneous tissue disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Angioedema (Skin and subcutaneous tissue disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Heat rash (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Keratosis pilaris (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Rash rubelliform (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Exposure to communicable disease (Social circumstances) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Haematoma (Vascular disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Tenderness (Any) (Skin and subcutaneous tissue disorders) | 192/264 | 195/270 | 0/0 | 0/0 | 121/149 | 124/147 | 0/0 | 0/0 — Infant Series Dose 1 and Toddler Dose; Tenderness (any)=present at site of vaccination.
Tenderness (Any) (Skin and subcutaneous tissue disorders) | 154/200 | 164/216 | 0/0 | 0/0 | 0/0 | 0/0 | 0/0 | 0/0 — Infant Series Dose 2; Tenderness (any)
Tenderness (Any) (Skin and subcutaneous tissue disorders) | 140/178 | 140/173 | 0/0 | 0/0 | 0/0 | 0/0 | 0/0 | 0/0 — Infant Series Dose 3; Tenderness (any)
Tenderness (Significant) (Skin and subcutaneous tissue disorders) | 25/182 | 18/195 | 0/0 | 0/0 | 10/65 | 6/49 | 0/0 | 0/0 — Infant Series Dose 1 and Toddler Dose; Tenderness (significant)=present and interfered with limb movement.
Tenderness (Significant) (Skin and subcutaneous tissue disorders) | 13/123 | 15/131 | 0/0 | 0/0 | 0/0 | 0/0 | 0/0 | 0/0 — Infant Series Dose 2; Tenderness (significant)
Tenderness (Significant) (Skin and subcutaneous tissue disorders) | 8/91 | 8/86 | 0/0 | 0/0 | 0/0 | 0/0 | 0/0 | 0/0 — Infant Series Dose 3; Tenderness (significant)
Induration (Any) (Skin and subcutaneous tissue disorders) | 55/201 | 51/216 | 0/0 | 0/0 | 40/91 | 37/73 | 0/0 | 0/0 — Infant Series Dose 1 and Toddler Dose; Induration (any)=present at site of vaccination.
Induration (Any) (Skin and subcutaneous tissue disorders) | 44/141 | 43/146 | 0/0 | 0/0 | 0/0 | 0/0 | 0/0 | 0/0 — Infant Series Dose 2; Induration (any)
Induration (Any) (Skin and subcutaneous tissue disorders) | 44/116 | 38/103 | 0/0 | 0/0 | 0/0 | 0/0 | 0/0 | 0/0 — Infant Series Dose 3; Induration (any)
Induration (Mild) (Skin and subcutaneous tissue disorders) | 46/199 | 45/212 | 0/0 | 0/0 | 39/90 | 33/71 | 0/0 | 0/0 — Infant Series Dose 1 and Toddler Dose; Induration (mild)=0.5 centimeters (cm) to 2.0 cm.
Induration (Mild) (Skin and subcutaneous tissue disorders) | 42/141 | 37/142 | 0/0 | 0/0 | 0/0 | 0/0 | 0/0 | 0/0 — Infant Series Dose 2; Induration (mild)
Induration (Mild) (Skin and subcutaneous tissue disorders) | 40/113 | 38/103 | 0/0 | 0/0 | 0/0 | 0/0 | 0/0 | 0/0 — Infant Series Dose 3; Induration (mild)
Induration (Moderate) (Skin and subcutaneous tissue disorders) | 12/176 | 10/193 | 0/0 | 0/0 | 10/68 | 7/49 | 0/0 | 0/0 — Infant Series Dose 1 and Toddler Dose; Induration
Induration (Moderate) (Skin and subcutaneous tissue disorders) | 6/118 | 9/126 | 0/0 | 0/0 | 0/0 | 0/0 | 0/0 | 0/0 — Infant Series Dose 2; Induration (moderate)
Induration (Moderate) (Skin and subcutaneous tissue disorders) | 6/91 | 5/82 | 0/0 | 0/0 | 0/0 | 0/0 | 0/0 | 0/0 (0) — Infant Series Dose 3; Induration (moderate)
Induration (Severe) (Skin and subcutaneous tissue disorders) | 0/173 | 0/187 | 0/0 | 0/0 | 0/59 | 0/44 | 0/0 | 0/0 — Infant Series Dose 1 and Toddler Dose; Induration (severe) >7.0 cm.
Induration (Severe) (Skin and subcutaneous tissue disorders) | 0/116 | 0/120 | 0/0 | 0/0 | 0/0 | 0/0 | 0/0 | 0/0 — Infant Series Dose 2; Induration (severe)
Induration (Severe) (Skin and subcutaneous tissue disorders) | 0/87 | 0/79 | 0/0 | 0/0 | 0/0 | 0/0 | 0/0 | 0/0 — Infant Series Dose 3; Induration (severe)
Erythema (Any) (Skin and subcutaneous tissue disorders) | 72/202 | 72/223 | 0/0 | 0/0 | 56/103 | 57/87 | 0/0 | 0/0 — Infant Series Dose 1 and Toddler Dose; Erythema (any)=present at site of vaccination.
Erythema (Any) (Skin and subcutaneous tissue disorders) | 70/155 | 62/164 | 0/0 | 0/0 | 0/0 | 0/0 | 0/0 | 0/0 — Infant Series Dose 2; Erythema (any)
Erythema (Any) (Skin and subcutaneous tissue disorders) | 64/131 | 59/118 | 0/0 | 0/0 | 0/0 | 0/0 | 0/0 | 0/0 — Infant Series Dose 3; Erythema (any)
Erythema (Mild) (Skin and subcutaneous tissue disorders) | 69/200 | 69/220 | 0/0 | 0/0 | 55/102 | 54/85 | 0/0 | 0/0 — Infant Series Dose 1 and Toddler Dose; Erythema (mild)=0.5 cm to 2.0 cm.
Erythema (Mild) (Skin and subcutaneous tissue disorders) | 69/155 | 60/162 | 0/0 | 0/0 | 0/0 | 0/0 | 0/0 | 0/0 — Infant Series Dose 2; Erythema (mild)
Erythema (Mild) (Skin and subcutaneous tissue disorders) | 61/128 | 57/117 | 0/0 | 0/0 | 0/0 | 0/0 | 0/0 | 0/0 — Infant Series Dose 3; Erythema (mild)
Erythema (Moderate) (Skin and subcutaneous tissue disorders) | 8/177 | 5/191 | 0/0 | 0/0 | 5/62 | 7/50 | 0/0 | 0/0 — Infant Series Dose 1 and Toddler Dose; Erythema (moderate)=2.5 cm to 7.0 cm.
Erythema (Moderate) (Skin and subcutaneous tissue disorders) | 2/117 | 4/124 | 0/0 | 0/0 | 0/0 | 0/0 | 0/0 | 0/0 — Infant Series Dose 2; Erythema (moderate)
Erythema (Moderate) (Skin and subcutaneous tissue disorders) | 5/91 | 4/80 | 0/0 | 0/0 | 0/0 | 0/0 | 0/0 | 0/0 — Infant Series Dose 3; Erythema (moderate)
Erythema (Severe) (Skin and subcutaneous tissue disorders) | 0/173 | 0/186 | 0/0 | 0/0 | 0/59 | 0/44 | 0/0 | 0/0 — Infant Series Dose 1 and Toddler Dose; Erythema (severe) >7.0 cm.
Erythema (Severe) (Skin and subcutaneous tissue disorders) | 0/116 | 0/120 | 0/0 | 0/0 | 0/0 | 0/0 | 0/0 | 0/0 — Infant Series Dose 2; Erythema (severe)
Erythema (Severe) (Skin and subcutaneous tissue disorders) | 0/87 | 0/79 | 0/0 | 0/0 | 0/0 | 0/0 | 0/0 | 0/0 — Infant Series Dose 3; Erythema (severe)
Fever ≥38°C but ≤39°C (General disorders) | 47/196 | 43/203 | 0/0 | 0/0 | 53/99 | 39/76 | 0/0 | 0/0 — Infant Series Dose 1 and Toddler Dose; Fever ≥38 degrees C but ≤39 degrees C
Fever ≥38°C but ≤39°C (General disorders) | 63/146 | 61/151 | 0/0 | 0/0 | 0/0 | 0/0 | 0/0 | 0/0 — Infant Series Dose 2; Fever ≥38 degrees C but ≤39 degrees C
Fever ≥38°C but ≤39°C (General disorders) | 49/123 | 40/106 | 0/0 | 0/0 | 0/0 | 0/0 | 0/0 | 0 — Infant Series Dose 3; Fever ≥38 degrees C but ≤39 degrees C
Fever >39°C but ≤40°C (General disorders) | 5/177 | 0/187 | 0/0 | 0/0 | 4/61 | 6/48 | 0/0 | 0/0 — Infant Series Dose 1 and Toddler Dose; Fever >39 degrees C but ≤40 degrees C
Fever >39°C but ≤40°C (Skin and subcutaneous tissue disorders) | 3/118 | 6/123 | 0/0 | 0/0 | 0/0 | 0/0 | 0/0 | 0/0 — Infant Series Dose 2; Fever >39 degrees C but ≤40 degrees C
Fever >39°C but ≤40°C (General disorders) | 8/94 | 2/81 | 0/0 | 0/0 | 0/0 | 0/0 | 0/0 | 0/0 — Infant Series Dose 3; Fever >39 degrees C but ≤40 degrees C
Fever >40°C (General disorders) | 0/174 | 0/187 | 0/0 | 0/0 | 1/60 | 0/45 | 0/0 | 0/0 — Infant Series Dose 1 and Toddler Dose; Fever >40 degrees C
Fever >40°C (General disorders) | 0/116 | 1/121 | 0/0 | 0/0 | 0/0 | 0/0 | 0/0 | 0/0 — Infant Series Dose 2; Fever >40 degrees C
Fever >40°C (General disorders) | 0/87 | 1/80 | 0/0 | 0/0 | 0/0 | 0/0 | 0/0 | 0/0 — Infant Series Dose 3; Fever >40 degrees C
Decreased appetite (General disorders) | 125/228 | 108/238 | 0/0 | 0/0 | 76/116 | 81/110 | 0/0 | 0/0 — Infant Series Dose 1 and Toddler Dose; Decreased appetite
Decreased appetite (General disorders) | 106/177 | 91/174 | 0/0 | 0/0 | 0/0 | 0/0 | 0/0 | 0/0 — Infant Series Dose 2; Decreased appetite
Decreased appetite (General disorders) | 87/147 | 81/136 | 0/0 | 0/0 | 0/0 | 0/0 | 0/0 | 0/0 — Infant Series Dose 3; Decreased appetite
Irritability (General disorders) | 259/289 | 249/290 | 0/0 | 0/0 | 183/199 | 163/175 | 0/0 | 0/0 — Infant Series Dose 1 and Toddler Dose; Irritability
Irritability (General disorders) | 212/236 | 216/236 | 0/0 | 0/0 | 0/0 | 0/0 | 0/0 | 0/0 — Infant Series Dose 2; Irritability
Irritability (General disorders) | 191/216 | 201/218 | 0/0 | 0/0 | 0/0 | 0/0 | 0/0 | 0/0 — Infant Series Dose 3; Irritability
Increased sleep (General disorders) | 213/268 | 212/270 | 0/0 | 0/0 | 81/115 | 81/109 | 0/0 | 0/0 — Infant Series Dose 1 and Toddler Dose; Increased sleep
Increased sleep (General disorders) | 161/203 | 147/200 | 0/0 | 0/0 | 0/0 | 0/0 | 0/0 | 0/0 — Infant Series Dose 2; Increased sleep
Increased sleep (General disorders) | 117/164 | 104/149 | 0/0 | 0/0 | 0/0 | 0/0 | 0/0 | 0/0 — Infant Series Dose 3; Increased sleep
Decreased sleep (General disorders) | 101/221 | 113/236 | 0/0 | 0/0 | 66/113 | 61/95 | 0/0 | 0/0 — Infant Series Dose 1 and Toddler Dose; Decreased sleep
Decreased sleep (General disorders) | 83/169 | 96/172 | 0/0 | 0/0 | 0/0 | 0/0 | 0/0 | 0/0 — Infant Series Dose 2; Decreased sleep
Decreased sleep (General disorders) | 93/154 | 85/134 | 0/0 | 0/0 | 0/0 | 0/0 | 0/0 | 0/0 — Infant Series Dose 3; Decreased sleep
Hives (urticaria) (General disorders) | 3/178 | 2/188 | 0/0 | 0/0 | 3/62 | 3/47 | 0/0 | 0/0 — Infant Series Dose 1 and Toddler Dose; Hives (urticaria)
Hives (urticaria) (General disorders) | 3/118 | 0/120 | 0/0 | 0/0 | 0/0 | 0/0 | 0/0 | 0/0 — Infant Series Dose 2; Hives (urticaria)
Hives (urticaria) (General disorders) | 4/89 | 0/79 | 0/0 | 0/0 | 0/0 | 0/0 | 0/0 | 0/0 — Infant Series Dose 3; Hives (urticaria)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Pfizer has the right to review disclosures, requesting a delay of less than 60 days. Investigator will postpone single center publications until after disclosure of pooled data (all sites), less than 12 months from study completion/termination at all participating sites. Investigator may not disclose previously undisclosed confidential information other than study results.